CLINICAL TRIAL: NCT01379690
Title: Association of HBA1C and Hip Fractures in Elderly Type 2 Diabetic Patients
Brief Title: Retrospective Study: Hip Fractures in Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Changi General Hospital (Other)
Responsible Party: Principal Investigator, Puar Hai Kiat Troy, Medical Doctor, Changi General Hospital
Other Study IDs: ChangiGH
Record Dates: First submitted 2011-06-22; First posted 2011-06-23 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2012-02

CONDITIONS: Type 2 Diabetes; Hip Fractures
Keywords: HbA1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hip Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: Controls were selected from patients with diabetes on consultation during the year 2005-2010 in specialist clinic, without a previous hip fracture. There was no followup period for these patients. Instead the A1C value upon the point of consultation was used to reflect glycaemic control at the point of consultation
  Interventions: Other: HBA1C
- Case: All patients with treated diabetes admitted with primary diagnosis hip fractures from 2005-2010 to Changi General Hospital was included in the study. The A1C at the point of admission was used to reflect the glycaemic control at that point in time. This was a retrospective study and there was no subsequent follow up on patients after the point of admission
  Interventions: Other: HBA1C

INTERVENTIONS:
Other: HBA1C — Used level of HBA1C as a reflection of glycaemic control of the cases and controls

SUMMARY:
Type 2 DM patients are at increased risk of falls as a consequence of long term hyperglycemic complications including retinopathy and neuropathy, and also as a result of hypoglycaemic therapy. Values of A1C <= 7% has been shown to increase the risk of falls in elderly T2DM patients .

Increased fall risk may explain why T2DM patients are at increased risk of hip fractures , despite having a higher bone mineral density as compared to non-T2DM patients. Given the high morbidity and mortality (25% mortality in 1st year post-fracture) associated with hip fractures , all care must be given to prevent hip fractures in T2DM patients.

There is controversial data on T2DM medications and fracture risk. Vestergaard showed that use of metformin and sulphonylureas decreased the risk of all fractures, while there was there was a similar trend with insulin.

The present study sought to evaluate the relationship between A1c values and the risk of fractures in treated patients with T2DM.

DETAILED DESCRIPTION:
This was a retrospective case-control study. All patients with T2DM admitted with a primary diagnosis of hip fracture and a A1c performed within 3 months of the event admitted to Changi General Hospital, Singapore from 1st Jan 2005 to 31st Dec 2010were included in the study. As the present study was targeted at looking at an association between the glucose lowering effect of medications on A1C levels and subsequent hip fracture risk, exclusion criteria included patients who wereduplicate cases, traumatic fractures, newly diagnosed T2DM patients, and those on diet control.

The information on discharge diagnosis was taken from the Discharge Register of the Hospital. It includes all diagnosis of the patient upon discharge. The diagnosis of patients is coded using the International Classification of Diseases (ICD) system. All patients admitted with the diagnosis of neck of femur fracture (8208 ICD-9), inter-trochanteric fracture (82021 ICD-9), sub-trochanteric fracture (82022 ICD-9), transcervical fracture (82003 ICD-9), and a secondary diagnosis of diabetes (250 ICD-9) were identified from the register.

Out of 932 patients initially identified, 31 were duplicates, 10 were admitted for a traumatic fracture, 136 had no recent A1C level. Of the remaining 757 patients, 162 on diet control and 12 newly diagnosed with diabetes were excluded. The final list of cases consisted of 581 patients, 157 men and 427 women, mean age 76.3 ± 8.7 years.

Controls were selected from a register of patients managed for diabetes from a similar period (1st Jan 2005 to 31st Dec 2010) at Changi General Hospital outpatient clinics (N=4,522). For each case, one control subject, matched for sex and within 2 years of age, was randomly selected from the register. Inclusion criteria included patients taking oral hypoglycemic agents or insulin, and exclusion criteria were patients with a history of hip fractures.

Information on the baseline characteristics and exposure variables were collected by the same methods in cases and control subjects, using the computerised medical records and discernment of the medical notes.

The study was performed in accordance with the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetic Patients
* Hip fracture (Case) or no hip fracture (control)

Exclusion Criteria:

* Traumatic fractures
* on diet control for diabetes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All diabetic patients on treatment with medications, seen at Changi General Hospital from 2005-2010
Sampling Method: Probability Sample
Enrollment: 1162 (Actual)
Dates: Start 2011-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Hip Fracture | 2005-2010
  Admission for hip fracture

CONTACTS AND LOCATIONS:
Overall Officials: Troy H Puar, MRCP, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Vestergaard P, Rejnmark L, Mosekilde L. Relative fracture risk in patients with diabetes mellitus, and the impact of insulin and oral antidiabetic medication on relative fracture risk. Diabetologia. 2005 Jul;48(7):1292-9. doi: 10.1007/s00125-005-1786-3. Epub 2005 May 21. PMID 15909154